CLINICAL TRIAL: NCT06063486
Title: A Phase 2, Double-blind, Randomized Study to Compare the Effect of Curcumin Versus Placebo on Inflammatory Cytokines, Symptoms and Disease Parameters in Clonal Cytopenia of Undetermined Significance (CCUS), Low-Risk Myelodysplastic Syndrome (LR-MDS), and Myeloproliferative Neoplasms (MPNs)
Brief Title: Curcumin to Improve Inflammation and Symptoms in Patients With Clonal Cytopenia of Undetermined Significance, Low Risk Myelodysplastic Syndrome, and Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9L-23-1; NCI-2023-06976 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-23-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-09-23; First posted 2023-10-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Clonal Cytopenia of Undetermined Significance; Essential Thrombocythemia; Myelodysplastic Syndrome; Myelofibrosis; Polycythemia Vera
MeSH Terms: conditions — Thrombocythemia, Essential; Myelodysplastic Syndromes; Primary Myelofibrosis; Polycythemia Vera | interventions — Specimen Handling; Biopsy; Curcumin; demethoxycurcumin; piperine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (C3 Complex/Bioperine) (Experimental): Patients receive C3 complex/Bioperine PO BID for 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy at baseline and follow up, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Dietary Supplement: Curcumin/ Demethoxycurcumin/Bisdemethoxycurcumin-containing Supplement; Dietary Supplement: Piperine Extract (Standardized); Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO BID for 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy at baseline and follow up, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Dietary Supplement: Curcumin/ Demethoxycurcumin/Bisdemethoxycurcumin-containing Supplement — Given PO
  Other Names: Curcumin C3 Complex
  Arms: Arm I (C3 Complex/Bioperine)
Dietary Supplement: Piperine Extract (Standardized) — Given PO
  Other Names: Bioperine; Standardized Piperine Extract
  Arms: Arm I (C3 Complex/Bioperine)
Drug: Placebo Administration — Given PO
  Other Names: Sugar pills
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial evaluates how a curcumin supplement (C3 complex/Bioperine) changes the inflammatory response and symptomatology in patients with clonal cytopenia of undetermined significance (CCUS), low risk myelodysplastic syndrome (LR-MDS), and myeloproliferative neoplasms (MPN). Chronic inflammation drives disease development and contributes to symptoms experienced by patients with CCUS, LR-MDS, and MPN. Curcumin has been shown to have anti-inflammatory and anti-cancer properties and has been studied in various chronic illnesses and hematologic diseases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the change in inflammatory cytokine levels in study patients treated with curcumin versus placebo over a 12-month follow-up period.

II. To compare the change in symptomatology in study patients treated with curcumin versus placebo over a 12-month follow-up period.

SECONDARY OBJECTIVES:

I. To investigate the effect on variant allele frequency (VAF) of baseline mutations in study patients treated with curcumin versus placebo.

II. To investigate the effect on methylation patterns in study patients treated with curcumin versus placebo.

III. To evaluate the effect on peripheral blood cells in study patients treated with curcumin versus placebo.

IV. To assess the safety of curcumin for patients with CCUS/LR-MDS and symptomatic MPN who do not require disease-modifying therapy.

EXPLORATORY OBJECTIVE:

I. To investigate the correlation between inflammatory cytokine levels and symptom scores in study patients treated with curcumin versus placebo.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: Patients receive curcumin/demethoxycurcumin/bisdemethoxycurcumin-containing supplement (C3 complex)/piperine extract (standardized) (Bioperine) orally (PO) twice daily (BID) for 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy at baseline and follow up, and collection of blood samples throughout the trial.

Arm II: Patients receive placebo PO BID for 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and biopsy at baseline and follow up, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Ability to understand and willingness to sign a written informed consent
* Diagnosis of polycythemia vera (PV), essential thrombocytosis (ET) or myelofibrosis (MF) per World Health Organization (WHO) 2016 diagnostic criteria

  * Presence of at least one symptom measurable using the MPN-/Symptom Assessment Form (SAF) with a severity greater than 3
  * MPN patients determined to have stable disease undergoing surveillance and unlikely to require initiation of new cytoreductive therapy (i.e., hydroxyurea, ruxotinib, interferon within the study period); patients on a stable dose of hydroxyurea for at least 6 months who meet the other inclusion/exclusion criteria may be included
* A diagnosis of CCUS or LR-MDS

  * CCUS defined as persistent cytopenia for > 6 months (hemoglobin [Hgb] < 11.3 g/dL [7 mmol/L] in women and Hgb < 12.9 g/dL [8 mmol/L] in men, platelet < 150 x 10^9/L or neutrophils < 1.8 x 10^9/L), normal cytogenetics, presence of detectable MDS associated mutations and bone marrow morphology non-diagnostic of MDS or any other malignancies
  * LR-MDS as defined by WHO 2016 diagnosis criteria
  * Minimum baseline symptom score of 25 in the fatigue section of the symptom questionnaire

Exclusion Criteria:

* Patients with intake of curcumin as a dietary supplement, including multivitamin and unwillingness to quit more than 24 hours before study start
* Patients with inability to understand and adhere to information given
* Patients receiving active treatment for another malignancy except with hormonal therapy for a malignancy considered to be in remission or growth factors (erythropoietin, granulocyte colony-stimulating factor [G-CSF] and luspatercept)
* Patients with intermediate or high-risk MDS
* Patients must not be pregnant or nursing
* Patients must not be on any oral or intravenous steroid or any other anti-inflammatories (ibuprofen > 200mg/week or 400mg/month, naproxen of any dose, > 325mg aspirin daily, any herbal anti-inflammatory concoction of any dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in peripheral blood levels of inflammatory cytokines | At baseline, 3 months, and 12 months
  Interleukin (IL) 1beta, IL-6, IL-18, transforming growth factor-beta, and tumor necrosis factor-alpha will be assessed. Mean inflammatory cytokine changes in the treatment group will be compared to that of the control group. A two-sided two-sample unequal-variance t-test will be applied to compare the difference of the mean of changes at 12-months from the baseline measurement between the two arms, respectively. P-values from the test and the 95% confidence interval of the estimated difference will be reported for each of the inflammatory cytokines.
Mean change in symptom scores for clonal cytopenia of undetermined significance and low risk myelodysplastic syndrome patients | At baseline, 3 months, 12 months
  Symptoms scores will be assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 version 3 (EORTC-QLQ-C30 version 3).This is a validated tool for assessing health-related quality of life in cancer patients. The questionnaire is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. Scores range from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.(no symptom) to 10 (worst possible symptom).
Mean change in symptom scores for myeloproliferative neoplasm (MPN) patients | At baseline, 3 months, 12 months
  MPN-related symptoms will be assessed using the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score. Possible scores range from 0 (no symptom) to 10 (worst possible symptom).

SECONDARY OUTCOMES:
Change in the variant allele frequency of mutated clones | After 12 months of treatment
  Both parametric methods i.e., the two-sample t-test and the non-parametric Wilcoxon rank sum test (with no assumption on the distribution of the data) will be applied.
Change in the deoxyribonucleic acid methylation pattern | After 12 months of treatment
  Both parametric methods i.e., the two-sample t-test and the non-parametric Wilcoxon rank sum test (with no assumption on the distribution of the data) will be applied.
Change in peripheral blood cell counts | After 12 months of treatment
  Peripheral blood cell counts will include absolute neutrophil count, hemoglobin, and platelets. Change in peripheral blood cell counts will be compared to pretreatment. Both parametric methods i.e., the two-sample t-test and the non-parametric Wilcoxon rank sum test (with no assumption on the distribution of the data) will be applied.
Safety of curcumin in patients with CCUS/LR-MDS and symptomatic MPN | Every 2 weeks for the first month of treatment, every month for the following 2 months, then every 3 months for a total of 12 months.
  Will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0.
Change in the rate of transfusion requirement measured | Up to 10 years
  Will be measured by the number of units required per 8-week period. Both parametric methods i.e., the two-sample t-test and the non-parametric Wilcoxon rank sum test (with no assumption on the distribution of the data) will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Casey L O'Connell, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California